CLINICAL TRIAL: NCT00990236
Title: Thrombelastography Based Dosing of Enoxaparin for Thromboprophylaxis: a Prospective Randomized Trial
Brief Title: Thrombelastography Based Dosing of Enoxaparin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Medical Research Foundation, Oregon (Other); National Trauma Research Institute (Other)
Responsible Party: Principal Investigator, Martin A Schreiber, MD, Professor & Chief of Trauma, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 001-01
Record Dates: First submitted 2009-09-29; First posted 2009-10-06 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Thromboembolic Complications
Keywords: deep vein thrombosis; superficial venous thrombosis; pulmonary embolus
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Enoxaparin; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enoxaparin 30 mg BID (Active Comparator): standard dose enoxaparin thromboprophylaxis (30 mg twice daily)
  Interventions: Drug: Enoxaparin 30 mg BID
- Enoxaparin dose adjusted based on TEG (Experimental): enoxaparin dose modified based on TEG results
  Interventions: Drug: Enoxaparin dose adjusted Lovenox based on TEG

INTERVENTIONS:
Drug: Enoxaparin dose adjusted Lovenox based on TEG — Enoxaparin doses will be adjusted (10 mg BID) based on delta-R results from TEG. Delta-R < 1.0 min - increase dose by 10 mg BID; delta-R >/= 1.0 min and </= 2.0 min - no change; delta-R > 2.0 min - decrease dose by 10 mg BID.
  Other Names: enoxaparin, lovenox
  Arms: Enoxaparin dose adjusted based on TEG
Drug: Enoxaparin 30 mg BID — Enoxaparin dose of 30 mg twice a day without any adjustments
  Other Names: enoxaparin, lovenox
  Arms: Enoxaparin 30 mg BID

SUMMARY:
The risk of developing a blood clot occurs in up to 60% of all critical care patients. Many times enoxaparin (or Lovenox®) is given to patients who are at a higher risk of developing clots in their legs or lungs. Recent data suggest that a standard dose of Lovenox may not fully prevent the development of these clots especially in critically ill or obese patients. Routine enoxaparin dosing can also result in bleeding complications. Thrombelastography (TEG®) can be used to measure how blood clots. The purposes of this study are:

* to learn if the TEG® can better guide physicians in prescribing an effective dose of Lovenox compared to standard doses recommended by the drug company in preventing blood clots from developing in the legs and lungs, and
* to compare the development of blood clots in patients receiving the standard dose of enoxaparin compared to patients receiving a TEG® guided dose of enoxaparin.
* to determine if TEG guided dosing results in decreased bleeding complications compared to standard dosing.

DETAILED DESCRIPTION:
Hypothesis:

Enoxaparin dosed to maintain a TEG® ΔR greater than 1.0 minute will decrease the incidence of DVT compared to standard dosing.

Initiation of enoxaparin thromboprophylaxis will be done by the treatment team. Once enrolled, the subject will be randomized to continue receiving standard dose enoxaparin (30 mg twice daily) or variable TEG® guided enoxaparin dosing. The treatment team and the subject will be blinded regarding the arm in which the patient is enrolled. Patient characteristics: age, gender, body mass index (BMI), comorbidities, Acute Physiology and Chronic Health Evaluation II score (APACHE II), injuries, and operations will be collected. As part of standard protocol in the ICU, all patients will undergo weekly ultrasound duplex examination of the lower extremities for presence of deep venous thrombosis.

A baseline TEG® will be completed on each patient when they are enrolled in the study. The blood will be drawn between four and six hours after the morning dose is administered, corresponding to maximum tissue levels of enoxaparin. TEG® assays will be run in duplicate for each patient, with and without heparinase, which negates the effects of enoxaparin in the assay.

Those patients randomized to the control arm of the study will have TEG® performed at baseline and daily for one week, then twice weekly. The twice weekly TEG® assays will be done until the patient is discharged from inpatient care or enoxaparin is discontinued by the treatment team. No adjustments will be made to their enoxaparin dosing.

Patients in the TEG® guided enoxaparin dosing arm will start treatment as ordered by the primary treatment team. After the second TEG®, the dose of enoxaparin will be adjusted in 10 mg increments per dose in order to reach a target ΔR between 1.0 and 1.4 minutes. If the initial ΔR is greater than 1.4 minutes, the dose of enoxaparin will be decreased by 10 mg increments until the target ΔR is achieved. Patients will have TEGs® performed daily and adjustment of dosing until the target ΔR is reached. Once the target ΔR is achieved, TEG® will be done twice weekly until the patient is discharged from inpatient care or enoxaparin is discontinued by the treatment team. All patients will be assessed daily by study personnel for bleeding complications. If bleeding complications occur, subjects will be withdrawn from the study. If interim analysis identifies a significant difference in bleeding complications between groups the study will be terminated.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient initiated on enoxaparin thromboprophylaxis
* Age greater than 15 years

Exclusion Criteria:

* Unable to obtain consent from patient or ARR
* Presence of: intracranial hemorrhage, brain injury
* Receiving therapeutic dose enoxaparin
* Receiving other forms of anticoagulation
* Receiving non-standard dosing regimen of enoxaparin

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2009-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schreiber, MD FACS, Principal Investigator — Oregon Health and Science University
Locations (3):
- United States (3):
  - Oregon Health & Science University, Portland, Oregon
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Connelly CR, Van PY, Hart KD, Louis SG, Fair KA, Erickson AS, Rick EA, Simeon EC, Bulger EM, Arbabi S, Holcomb JB, Moore LJ, Schreiber MA. Thrombelastography-Based Dosing of Enoxaparin for Thromboprophylaxis in Trauma and Surgical Patients: A Randomized Clinical Trial. JAMA Surg. 2016 Oct 19;151(10):e162069. doi: 10.1001/jamasurg.2016.2069. Epub 2016 Oct 19. PMID 27487253

RESULTS

PARTICIPANT FLOW:
Groups:
- Exoxaparin 30 mg BID: standard dose enoxaparin thromboprophylaxis (30 mg twice daily)
  Dose-adjusted Lovenox based on TEG: Lovenox doses will be adjusted (10 mg BID) based on delta-R results from TEG. Delta-R < 1.0 min - increase dose by 10 mg BID; delta-R >/= 1.0 min and </= 2.0 min - no change; delta-R > 2.0 min - decrease dose by 10 mg BID.
- Enoxaparin Dose Adjusted Based on TEG: enoxaparin dose modified based on TEG results
  Dose-adjusted Lovenox based on TEG: Lovenox doses will be adjusted (10 mg BID) based on delta-R results from TEG. Delta-R < 1.0 min - increase dose by 10 mg BID; delta-R >/= 1.0 min and </= 2.0 min - no change; delta-R > 2.0 min - decrease dose by 10 mg BID.
Period: Overall Study
Arm/Group | Exoxaparin 30 mg BID | Enoxaparin Dose Adjusted Based on TEG
Started | 89 | 96
Completed | 89 | 96
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exoxaparin 30 mg BID | Enoxaparin Dose Adjusted Based on TEG | Total
Number analyzed (Participants) | 89 | 96 | 185
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44.0 [28.0 to 60.0] | 48.5 [33.8 to 58.2] | 46.0 [32.0 to 59.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 25 | 65
  Male | 49 | 71 | 120
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 89 | 96 | 185

OUTCOME MEASURES:

1. Primary Outcome: Development of Deep Vein Thrombosis (DVT)
Description: An ultrasound duplex will be completed at least one time after randomization to determine if the subject has developed a DVT.
Time Frame: Through study completion, assessed up to 120 days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Exoxaparin 30 mg BID | Enoxaparin Dose Adjusted Based on TEG
Number analyzed (Participants) | 89 | 96
Participants | 6 | 5

2. Secondary Outcome: Incidence of Bleeding Complications
Description: An increase in bleeding complications will be assessed daily during hospitalization
Time Frame: Through study completion, assessed up to 120 days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Exoxaparin 30 mg BID | Enoxaparin Dose Adjusted Based on TEG
Number analyzed (Participants) | 89 | 96
Participants | 5 | 13

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for a period up to 120 days.
Arm/Group | Exoxaparin 30 mg BID | Enoxaparin Dose Adjusted Based on TEG
All-Cause Mortality (participants affected / at risk) | 0/89 | 2/96
Serious Adverse Events (participants affected / at risk) | 0/89 | 1/96
Other Adverse Events (participants affected / at risk) | 1/89 | 1/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exoxaparin 30 mg BID (N=89) | Enoxaparin Dose Adjusted Based on TEG (N=96)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exoxaparin 30 mg BID (N=89) | Enoxaparin Dose Adjusted Based on TEG (N=96)
Superficial venous thrombosis (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No